CLINICAL TRIAL: NCT03106584
Title: Investigating the Potential for Marigot's Nutrition Supplement to Improve Symptoms and Physical Function in Those With Mild to Moderate Knee Osteoarthritis (KOA) Versus the Current Market Leader (Glucosamine Sulphate)
Brief Title: The Marigot Osteoarthritis Nutritional Intervention (MOANi) Trial
Acronym: MOANi
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University College Dublin (Other)
Collaborators: Marigot Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LS-17-10-Delahunt-DeVito
Record Dates: First submitted 2017-03-22; First posted 2017-04-10 (Actual); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Knee Osteoarthritis
Keywords: Knee pain; Glucosamine; WOMAC; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Glucosamine

STUDY DESIGN:
Intervention Model Description: The project is a double blind randomized controlled clinical trial (pilot), with a cross-over design. Participants, will be randomized to begin taking either Aquamin-plus or Glucosamine sulphate following medical diagnosis and baseline assessment.
  Following 12 weeks of supplementation of Glucosamine sulphate or Aquamin-plus there will be a 4-week washout period before participants consume the other supplement.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The supplements provided by Marigot Ltd. will be marked either A or B. No member of the research team will be aware of the ingredients in either of the supplements, the only distinguishing feature will be the labels - A and B. It is for this reason that we can say that the study will be double blind as neither investigators nor participants will have any knowledge of the supplement that they will be consuming.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glucosamine sulphate (Active Comparator): Glucosamine sulphate will be consumed as either supplement A or B (i.e. blinded) for a period of 12-weeks. Glucosamine will be taken 2 times daily with food.
  After 12 weeks of supplementation, participants will begin taking the alternative supplement (Aquamin-plus), after a washout period of not less than 1 month between the intervention arms of the study.
  Interventions: Dietary Supplement: Aquamin-Plus; Dietary Supplement: Glucosamine sulphate
- Aquamin-plus (Experimental): Aquamin-plus will be consumed as either supplement A or B (i.e. blinded) for a period of 12-weeks. Aquamin-plus will be taken 2 times daily with food.
  After 12 weeks of supplementation, participants will begin taking the alternative supplement (Glucosamine sulphate), after a washout period of not less than 1 month between the intervention arms of the study.
  Interventions: Dietary Supplement: Aquamin-Plus; Dietary Supplement: Glucosamine sulphate

INTERVENTIONS:
Dietary Supplement: Aquamin-Plus — Aquamin (a calcium-rich marine multi-mineral) - 666.7mg magnesium hydroxide - 66.66mg pine bark - 30mg vitamin d3 - 2.5μg
  Dosage:
  4 Capsules is equal to effective dose
Dietary Supplement: Glucosamine sulphate — The Glucosamine sulphate supplement contains 500mg of the active ingredient Glucosamine sulphate per serving (one capsule).
  Dosage:
  4 Capsules is equal to effective dose

SUMMARY:
The purpose of the study is to test 30 individuals with mild-moderate knee joint osteoarthritis to investigate whether the combination of Aquamin (a calcium-rich marine multi-mineral) and a polyphenol-rich pine bark extract (Enzogenol), when taken as a food supplement for 3 months has comparable or superior benefits to glucosamine sulphate in patients with painful knee osteoarthritis (KOA). From here on in we refer to Aquamin's combination product as Aquamin-plus. The main outcome measure is a reduction in pain.

Provision of data that demonstrate preliminary equivalency or superiority to current, non-pharmaceutical options such as glucosamine will broaden consumer choice, and provide them with an option that is supported by science, rather than marketing alone.

The hypothesis of the study is that the consumption of Aquamin-plus will have comparable effects on reducing pain in individuals with Knee Joint OA to glucosamine.

DETAILED DESCRIPTION:
This project will be a double blinded randomized cross-over control (pilot) trial that will investigate whether the combination of Aquamin (a calcium-rich marine multi-mineral) and a polyphenol-rich pine bark extract (Enzogenol), when taken as a food supplement for 3 months (12 weeks) has comparable or superior benefits to glucosamine sulphate in patients with painful knee osteoarthritis (KOA). From here on in we refer to Aquamin's combination product as Aquamin-plus. The main outcome measure is a reduction in pain (WOMAC index) and improve physical function (6MWD and TUG).

The hypothesis of the study is that the consumption of Aquamin-plus for a period of 3 months will have comparable or superior effects on to glucosamine sulphate in reducing pain and improving physical function in individuals with KOA.

According to the Food and Drug Administration et al. osteoarthritis (OA) can be defined as a serious disease or condition because, among other aspects, it is "…associated with morbidity that has substantial impact on day-to-day functioning…" . Furthermore, the current Osteoarthritis Research Society International (OARSI) definition of OA has been proposed as, "OA is a disorder involving movable joints characterized by cell stress and extracellular matrix degradation initiated by micro- and macro-injury that activates maladaptive repair responses including pro-inflammatory pathways of innate immunity. The disease manifests first as a molecular derangement (abnormal joint tissue metabolism) followed by anatomic, and/or physiologic derangements (characterized by cartilage degradation, bone remodeling, osteophyte formation, joint inflammation and loss of normal joint function), that can culminate in illness"

The condition can be characterized as a branch of rheumatic disease that is a progressive condition of synovial joints and is caused by the failure of a joint to repair following damage. This damage may have been caused by stresses due to an abnormality in the articular cartilage, subchondral bone, ligaments, menisci, periarticular muscles, peripheral nerves or synovium. Failure of these normal biological processes leads to breakdown of cartilage and bone and is characterized by symptoms of pain, stiffness, functional disability and can and lead to negative effects on fatigue, mood, sleep and overall quality of life. OA has the highest frequency of all rheumatic diseases and is one of the most prevalent chronic diseases in the modern day. According to the Global Burden of Disease (GBD) study, progressive ageing of the population could make OA the ninth cause of disability-adjusted life years (DALYs) in developed countries by the year 2020, with KOA accounting for 83% of the total OA burden.

Investigations into the heritability of OA have identified some interesting results. In a British twin cohort, the genetic contribution to radiographically defined hip and KOA was estimated to 39-65% in women with a Danish twin studies finding similar variance in hip arthroplasty due to OA (47%) but only 18% for knee arthroplasty due to OA. However, more recent data from a larger cohort (n = 9058) showed a heritability of 73% and 45% in hip and knee arthroplasty, respectively. Interestingly, identified that while hip OA associated arthroplasty remains highly heritable regardless of environmental factors, while the genetic component of KOA (for arthroplasty) was significantly modifiable with increasing BMI. These data show the requirement for clinical interventions to focus on symptomatic KOA, particularly considering the exponentially increasing BMI and obesity in the western world.

Data from The Irish Longitudinal Study on Ageing (TILDA) show that approximately 13% (women-17.3%, men-9.4%; self-reported) of Irish residence over the age of 50 suffer from symptomatic OA, with 19.2% of those reporting symptomatic KOA. These are similar to data from Arthritis Research UK showing an 18% prevalence of patients visiting a general practitioner presenting with symptoms of KOA. Moreover, these reported incidence rates are estimated to raise in tandem with population age (Arthritis Research UK, 2013). In fact, the prevalence of KOA in the US is 25% and increases by 2% each year, likely due to the aging population (as in the UK) and raising obesity rate, with a lifetime risk of symptomatic KOA as high as 60.5 % in obese individuals.

Joint pain is the most common complaint among those who seek medical care for OA and as a result of OA pain 80% of individuals with have some degree of movement limitation, 25% cannot perform major activities of daily living and 11% of adults with KOA need help with personal care. Consequentially, OA can lead to negative effects on quality of life, mood, fatigue and sleep. Interestingly, poor sleep occurs in ~70% of older individuals with OA and is linked with fatigue, which in turn is associated with a greater fall risk in the elderly and identifies fatigue as a further concern, in addition to joint instability, of fall-related complications.

OA is a progressive condition with no cure, however treatments do exist aimed at reducing symptoms and slowing progression of the disease. This in turn will improve mobility, quality of life and leads to a reduction in the need joint replacement surgery in the long-term and consequently reduces the demand on healthcare resource. Non-steroidal anti-inflammatory drugs (NSAID) are the traditional approach for clinical management of mild-to-moderate OA symptoms, however NSAIDs have been associated with potentially harmful side effects such as gastrointestinal complications, renal disturbances and cardiovascular events. Therefore, non-pharmaceutical alternatives have been developed such as glucosamine compounds, however the reported efficacy for reducing OA symptoms varies. Nonetheless, while glucosamine compounds have a lower risk of adverse effects compared to NSAIDs and other symptomatic slow-acting drugs for OA (SYSADOA), glucosamine compounds show higher risk of adverse side effects than placebo and as such alternatives should be sought. Further to possible adverse health effects, NSAIDs and SYASDOAs are costly and greatly affect the socioeconomic health of patients with OA. A recent meta-analysis of global generalized OA has shown that the individual annual incremental healthcare costs ranged from €705 to €19,715 and concluded that the social cost of OA could be between 0.25% and 0.50% of a country's GDP. More specifically, the individual cost of KOA (both social healthcare and private) can range from €528 to €11293 depending of severity. In fact, Hunter et al. recently called for urgent action to focus attention on opportunities to reduce the individual and socioeconomic burden of OA.

Glucosamine supplementation for the treatment of OA and OA related phenotypes spans many decades, with the first (to the authors' knowledge) patent filled in 1969 and research on human derived glucosamine published long before. The earliest identifiable mention (to the authors' knowledge) of Aqumin is from the late 90's with a patent, containing Aqumin, filled for human consumption in 2003, "Algae-based food supplement". Therefore, there is a significant advantage for glucosamine in the accumulation of large high quality studies into its therapeutic effects. Nonetheless, the few small pilot studies concerned with the therapeutic effects of Aquamin supplementation show promising results in comparison to both placebo and Glucosamine formulas. In fact, for some important OA phenotypes, Aquamin performs better, particularly in the reduction of NSAID use. While the proposed mechanisms of action differ considerable between the two supplements, inflammatory reduction occurs because of both. Currently, there have been no long-term trials concerned with the efficacy of Aquamin in the reduction of KOA related joint structural decline however, because Aquamin reduces inflammatory markers of KOA, albeit in only one small human study, it is possible that Aquamin might improve joint structural decline and KOA prognosis through possibly reducing joint tissue damage.

This project will be a double blinded randomized cross-over control trial with a sample size of 30 participants (based off a sample size calculation detailed below). The project will investigate two supplements on their effects on self-reported pain, quality of life, knee extensor/flexor strength, knee extensor/flexor myoelectric activity, functional mobility and biomarkers associated with inflammation. The participants will first be assessed for baseline measurements of the outcome measures mentioned above. They will then be randomly allocated to either group A or B and will take either supplement A or B for a period of 12 weeks. Following this there will be follow up assessments of the same outcome measures. This will be followed by a 4-week washout period prior to each subjects' baseline measures being reassessed and each participant allocated the 'other' supplement. After 12 weeks' supplementation, the subjects will then be retested for a final time.

An a priori sample size calculation indicated a total of 29 patients was required to enter this two-treatment crossover study to assess the primary outcomes. The probability is 80 percent that the study will detect a treatment difference at a two-sided 0.05 significance level, if the true difference between treatments is 12.000 units. This is based on the assumption that the within-patient standard deviation of the response variable is 15.62."

ELIGIBILITY:
Inclusion Criteria:

The project will focus on patients with a diagnosis of a mild-moderate KOA (level 1-3 Kellgren and Lawrence and WOMAC in the lower two quartiles), in the target knee, (Frestedt et al., 2008) and a BMI between 20 and 30 kg/m2.

Exclusion Criteria:

[1] rheumatoid arthritis [2] gout [3] pseudo gout [4] Paget's disease [5] seizure disorder [6] insulin dependent diabetes mellitus [7] uncontrolled hypertension [8] unstable cardiovascular disease [9] active hepatic or renal disease [10] active cancer and/or HIV infection, involved in other clinical trial or experimental treatments in the past 3 months; pregnant, lactating, or at risk of becoming pregnant; intramuscular/systemic corticosteroid injection within 4 weeks; intra-articular corticosteroid injection within 2 months; or inter-articular hyaluronic acid injection within 4 months prior to enrollment.

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-05-01 (Estimated); Primary Completion 2017-08-31 (Estimated); Study Completion 2017-10-01 (Estimated)

PRIMARY OUTCOMES:
Self reported KOA pain | Baseline, mid intervention (4 and 8 weeks) post intervention (12 weeks), post washout period (16 weeks), mid intervention (20 and 24 weeks) post intervention (28 weeks)
  The primary outcome measure will be an assessment of the participants' knee pain. This will be measured using the validated Western Ontario and McMaster Universities Arthritis Index (WOMAC) pain and function sub-scale. This will allow for the determination of the comparability, superiority or otherwise of Aquamin-plus compared to glucosamine sulphate in improving participant's self-reported knee pain and function. Change from baseline assessed.

SECONDARY OUTCOMES:
Quality of life questionnaire | Participants will be assessed on 4 separate occasions: Baseline, post intervention (12 weeks), post washout period (16 weeks), post intervention (28 weeks)
  This will be quantified by the EuroQoL-5D. The EuroQoL-5D will assess participants on their levels of function surrounding mobility, self-care, usual activities, pain / discomfort, anxiety / depression. Change from baseline assessed.
Knee flexor and extensor muscle strength | Participants will be assessed on 4 separate occasions: Baseline, post intervention (12 weeks), post washout period (16 weeks), post intervention (28 weeks)
  Participants knee joint strength will be assessed using an isokinetic dynamometer (Cybex). Specifically isometric strength of the quadricep and hamstring muscles. Change from baseline assessed.
Knee flexor and extensor muscle electrical activity | Participants will be assessed on 4 separate occasions: Baseline, post intervention (12 weeks), post washout period (16 weeks), post intervention (28 weeks)
  Muscles activation (via electromyography) during the performance of the isometric testing will be assessed for the quadricep and hamstring muscles. Both the agonist and antagonist muscle activity will be assessed and a co-contraction value will be calculated. Change from baseline assessed.
Biomarkers | Participants will be assessed on 4 separate occasions: Baseline, post intervention (12 weeks), post washout period (16 weeks), post intervention (28 weeks)
  Biomarkers known to be involved in the biological response to KOA will be assessed to investigate possible mechanistic effects and differences of both interventions. As such, in order to investigate these possible mechanistic parameters include venous blood sampling (10 mL). Change from baseline assessed.
Functional mobility | Participants will be assessed on 4 separate occasions: Baseline, post intervention (12 weeks), post washout period (16 weeks), post intervention (28 weeks)
  This will be assessed using the Six-minute Walk Test (6MWT) and the Timed Up and Go Test (TUG). These tests indicate levels of functional. Change from baseline assessed.
Body Composition | Participants will be assessed on 4 separate occasions: Baseline, post intervention (12 weeks), post washout period (16 weeks), post intervention (28 weeks)
  A Dule-Energy X ray Absorptimetry (DEXA) will be used to assess participants body composition. Change from baseline assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe De Vito, Prof., Study Chair — UCD; Eamonn Delahunt, PhD, Principal Investigator — UCD; Conor McCarthy, MD, Principal Investigator — Mater Misericordiae University Hospital
Locations (1):
- Institue for Sport and Health UCD, Dublin, Leinster, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Frestedt JL, Walsh M, Kuskowski MA, Zenk JL. A natural mineral supplement provides relief from knee osteoarthritis symptoms: a randomized controlled pilot trial. Nutr J. 2008 Feb 17;7:9. doi: 10.1186/1475-2891-7-9. PMID 18279523
- [Background] Frestedt JL, Kuskowski MA, Zenk JL. A natural seaweed derived mineral supplement (Aquamin F) for knee osteoarthritis: a randomised, placebo controlled pilot study. Nutr J. 2009 Feb 2;8:7. doi: 10.1186/1475-2891-8-7. PMID 19187557
- [Background] Murphy, C. T., et al.
- [Background] Kraus VB, Blanco FJ, Englund M, Karsdal MA, Lohmander LS. Call for standardized definitions of osteoarthritis and risk stratification for clinical trials and clinical use. Osteoarthritis Cartilage. 2015 Aug;23(8):1233-41. doi: 10.1016/j.joca.2015.03.036. Epub 2015 Apr 9. PMID 25865392
- [Background] Lane NE, Brandt K, Hawker G, Peeva E, Schreyer E, Tsuji W, Hochberg MC. OARSI-FDA initiative: defining the disease state of osteoarthritis. Osteoarthritis Cartilage. 2011 May;19(5):478-82. doi: 10.1016/j.joca.2010.09.013. Epub 2011 Mar 23. PMID 21396464
- [Background] Pena Ayala AH, Fernandez-Lopez JC. [Prevalence and risk factors in osteoarthritis]. Reumatol Clin. 2007 Oct;3 Suppl 3:S6-S12. doi: 10.1016/S1699-258X(07)73648-3. Epub 2008 Nov 13. Spanish. PMID 21794484
- [Background] Murphy L, Schwartz TA, Helmick CG, Renner JB, Tudor G, Koch G, Dragomir A, Kalsbeek WD, Luta G, Jordan JM. Lifetime risk of symptomatic knee osteoarthritis. Arthritis Rheum. 2008 Sep 15;59(9):1207-13. doi: 10.1002/art.24021. PMID 18759314
- [Background] Haq SA, Davatchi F. Osteoarthritis of the knees in the COPCORD world. Int J Rheum Dis. 2011 May;14(2):122-9. doi: 10.1111/j.1756-185X.2011.01615.x. PMID 21518310
- [Background] Lawrence RC, Felson DT, Helmick CG, Arnold LM, Choi H, Deyo RA, Gabriel S, Hirsch R, Hochberg MC, Hunder GG, Jordan JM, Katz JN, Kremers HM, Wolfe F; National Arthritis Data Workgroup. Estimates of the prevalence of arthritis and other rheumatic conditions in the United States. Part II. Arthritis Rheum. 2008 Jan;58(1):26-35. doi: 10.1002/art.23176. PMID 18163497
- [Background] Carmona L, Ballina J, Gabriel R, Laffon A; EPISER Study Group. The burden of musculoskeletal diseases in the general population of Spain: results from a national survey. Ann Rheum Dis. 2001 Nov;60(11):1040-5. doi: 10.1136/ard.60.11.1040. PMID 11602475
- [Background] Haugen IK, Englund M, Aliabadi P, Niu J, Clancy M, Kvien TK, Felson DT. Prevalence, incidence and progression of hand osteoarthritis in the general population: the Framingham Osteoarthritis Study. Ann Rheum Dis. 2011 Sep;70(9):1581-6. doi: 10.1136/ard.2011.150078. Epub 2011 May 27. PMID 21622766
- [Background] Hunter DJ, Schofield D, Callander E. The individual and socioeconomic impact of osteoarthritis. Nat Rev Rheumatol. 2014 Jul;10(7):437-41. doi: 10.1038/nrrheum.2014.44. Epub 2014 Mar 25. PMID 24662640
- [Background] Kopec JA, Richardson CG, Llewellyn-Thomas H, Klinkhoff A, Carswell A, Chalmers A. Probabilistic threshold technique showed that patients' preferences for specific trade-offs between pain relief and each side effect of treatment in osteoarthritis varied. J Clin Epidemiol. 2007 Sep;60(9):929-38. doi: 10.1016/j.jclinepi.2007.01.001. Epub 2007 May 8. PMID 17689809
- [Background] Magnusson K, Scurrah K, Ystrom E, Orstavik RE, Nilsen T, Steingrimsdottir OA, Ferreira P, Fenstad AM, Furnes O, Hagen KB. Genetic factors contribute more to hip than knee surgery due to osteoarthritis - a population-based twin registry study of joint arthroplasty. Osteoarthritis Cartilage. 2017 Jun;25(6):878-884. doi: 10.1016/j.joca.2016.12.015. Epub 2016 Dec 13. PMID 27986619
- [Background] Ng M, Fleming T, Robinson M, Thomson B, Graetz N, Margono C, Mullany EC, Biryukov S, Abbafati C, Abera SF, Abraham JP, Abu-Rmeileh NM, Achoki T, AlBuhairan FS, Alemu ZA, Alfonso R, Ali MK, Ali R, Guzman NA, Ammar W, Anwari P, Banerjee A, Barquera S, Basu S, Bennett DA, Bhutta Z, Blore J, Cabral N, Nonato IC, Chang JC, Chowdhury R, Courville KJ, Criqui MH, Cundiff DK, Dabhadkar KC, Dandona L, Davis A, Dayama A, Dharmaratne SD, Ding EL, Durrani AM, Esteghamati A, Farzadfar F, Fay DF, Feigin VL, Flaxman A, Forouzanfar MH, Goto A, Green MA, Gupta R, Hafezi-Nejad N, Hankey GJ, Harewood HC, Havmoeller R, Hay S, Hernandez L, Husseini A, Idrisov BT, Ikeda N, Islami F, Jahangir E, Jassal SK, Jee SH, Jeffreys M, Jonas JB, Kabagambe EK, Khalifa SE, Kengne AP, Khader YS, Khang YH, Kim D, Kimokoti RW, Kinge JM, Kokubo Y, Kosen S, Kwan G, Lai T, Leinsalu M, Li Y, Liang X, Liu S, Logroscino G, Lotufo PA, Lu Y, Ma J, Mainoo NK, Mensah GA, Merriman TR, Mokdad AH, Moschandreas J, Naghavi M, Naheed A, Nand D, Narayan KM, Nelson EL, Neuhouser ML, Nisar MI, Ohkubo T, Oti SO, Pedroza A, Prabhakaran D, Roy N, Sampson U, Seo H, Sepanlou SG, Shibuya K, Shiri R, Shiue I, Singh GM, Singh JA, Skirbekk V, Stapelberg NJ, Sturua L, Sykes BL, Tobias M, Tran BX, Trasande L, Toyoshima H, van de Vijver S, Vasankari TJ, Veerman JL, Velasquez-Melendez G, Vlassov VV, Vollset SE, Vos T, Wang C, Wang X, Weiderpass E, Werdecker A, Wright JL, Yang YC, Yatsuya H, Yoon J, Yoon SJ, Zhao Y, Zhou M, Zhu S, Lopez AD, Murray CJ, Gakidou E. Global, regional, and national prevalence of overweight and obesity in children and adults during 1980-2013: a systematic analysis for the Global Burden of Disease Study 2013. Lancet. 2014 Aug 30;384(9945):766-81. doi: 10.1016/S0140-6736(14)60460-8. Epub 2014 May 29. PMID 24880830
- [Background] French HP, Galvin R, Horgan NF, Kenny RA. Prevalence and burden of osteoarthritis amongst older people in Ireland: findings from The Irish LongituDinal Study on Ageing (TILDA). Eur J Public Health. 2016 Feb;26(1):192-8. doi: 10.1093/eurpub/ckv109. Epub 2015 Jun 23. PMID 26105959
- [Background] Murphy LB, Helmick CG, Schwartz TA, Renner JB, Tudor G, Koch GG, Dragomir AD, Kalsbeek WD, Luta G, Jordan JM. One in four people may develop symptomatic hip osteoarthritis in his or her lifetime. Osteoarthritis Cartilage. 2010 Nov;18(11):1372-9. doi: 10.1016/j.joca.2010.08.005. Epub 2010 Aug 14. PMID 20713163
- [Background] Blalock D, Miller A, Tilley M, Wang J. Joint instability and osteoarthritis. Clin Med Insights Arthritis Musculoskelet Disord. 2015 Feb 19;8:15-23. doi: 10.4137/CMAMD.S22147. eCollection 2015. PMID 25741184
- [Background] Reginster JY, Cooper C, Bruyere O. Re: Kucharz EJ, Kovalenko V, Szanto S, et al. A review of glucosamine for knee osteoarthritis: why patented crystalline glucosamine sulfate should be differentiated from other glucosamines to maximize clinical outcomes. Curr Med Res Opin 2016;32:997-1004. Curr Med Res Opin. 2016 Nov;32(11):1771-1772. doi: 10.1080/03007995.2016.1239575. Epub 2016 Sep 29. No abstract available. PMID 27649741
- [Background] Harirforoosh S, Asghar W, Jamali F. Adverse effects of nonsteroidal antiinflammatory drugs: an update of gastrointestinal, cardiovascular and renal complications. J Pharm Pharm Sci. 2013;16(5):821-47. doi: 10.18433/j3vw2f. PMID 24393558
- [Background] Richy F, Bruyere O, Ethgen O, Cucherat M, Henrotin Y, Reginster JY. Structural and symptomatic efficacy of glucosamine and chondroitin in knee osteoarthritis: a comprehensive meta-analysis. Arch Intern Med. 2003 Jul 14;163(13):1514-22. doi: 10.1001/archinte.163.13.1514. PMID 12860572
- [Background] McAlindon TE, LaValley MP, Gulin JP, Felson DT. Glucosamine and chondroitin for treatment of osteoarthritis: a systematic quality assessment and meta-analysis. JAMA. 2000 Mar 15;283(11):1469-75. doi: 10.1001/jama.283.11.1469. PMID 10732937
- [Background] Lee YH, Woo JH, Choi SJ, Ji JD, Song GG. Effect of glucosamine or chondroitin sulfate on the osteoarthritis progression: a meta-analysis. Rheumatol Int. 2010 Jan;30(3):357-63. doi: 10.1007/s00296-009-0969-5. Epub 2009 Jun 21. PMID 19544061
- [Background] Wandel S, Juni P, Tendal B, Nuesch E, Villiger PM, Welton NJ, Reichenbach S, Trelle S. Effects of glucosamine, chondroitin, or placebo in patients with osteoarthritis of hip or knee: network meta-analysis. BMJ. 2010 Sep 16;341:c4675. doi: 10.1136/bmj.c4675. PMID 20847017
- [Background] Murphy LB, Moss S, Do BT, Helmick CG, Schwartz TA, Barbour KE, Renner J, Kalsbeek W, Jordan JM. Annual Incidence of Knee Symptoms and Four Knee Osteoarthritis Outcomes in the Johnston County Osteoarthritis Project. Arthritis Care Res (Hoboken). 2016 Jan;68(1):55-65. doi: 10.1002/acr.22641. PMID 26097226
- [Background] Kongtharvonskul J, Anothaisintawee T, McEvoy M, Attia J, Woratanarat P, Thakkinstian A. Efficacy and safety of glucosamine, diacerein, and NSAIDs in osteoarthritis knee: a systematic review and network meta-analysis. Eur J Med Res. 2015 Mar 13;20(1):24. doi: 10.1186/s40001-015-0115-7. PMID 25889669
- [Background] Prieto-Alhambra D, Judge A, Javaid MK, Cooper C, Diez-Perez A, Arden NK. Incidence and risk factors for clinically diagnosed knee, hip and hand osteoarthritis: influences of age, gender and osteoarthritis affecting other joints. Ann Rheum Dis. 2014 Sep;73(9):1659-64. doi: 10.1136/annrheumdis-2013-203355. Epub 2013 Jun 6. PMID 23744977
- [Background] Oliveria SA, Felson DT, Reed JI, Cirillo PA, Walker AM. Incidence of symptomatic hand, hip, and knee osteoarthritis among patients in a health maintenance organization. Arthritis Rheum. 1995 Aug;38(8):1134-41. doi: 10.1002/art.1780380817. PMID 7639811
- [Background] Neogi T, Zhang Y. Epidemiology of osteoarthritis. Rheum Dis Clin North Am. 2013 Feb;39(1):1-19. doi: 10.1016/j.rdc.2012.10.004. Epub 2012 Nov 10. PMID 23312408
- [Background] Gabriel SE, Michaud K. Epidemiological studies in incidence, prevalence, mortality, and comorbidity of the rheumatic diseases. Arthritis Res Ther. 2009;11(3):229. doi: 10.1186/ar2669. Epub 2009 May 19. PMID 19519924
- [Background] Irvine, James Colquhoun, David McNicoll, and Alexander Hynd.
- [Background] MacGregor AJ, Antoniades L, Matson M, Andrew T, Spector TD. The genetic contribution to radiographic hip osteoarthritis in women: results of a classic twin study. Arthritis Rheum. 2000 Nov;43(11):2410-6. doi: 10.1002/1529-0131(200011)43:113.0.CO;2-E. PMID 11083262
- [Background] Spector TD, Cicuttini F, Baker J, Loughlin J, Hart D. Genetic influences on osteoarthritis in women: a twin study. BMJ. 1996 Apr 13;312(7036):940-3. doi: 10.1136/bmj.312.7036.940. PMID 8616305
- [Background] MacGregor AJ, Li Q, Spector TD, Williams FM. The genetic influence on radiographic osteoarthritis is site specific at the hand, hip and knee. Rheumatology (Oxford). 2009 Mar;48(3):277-80. doi: 10.1093/rheumatology/ken475. Epub 2009 Jan 19. PMID 19153142
- [Background] Skousgaard SG, Skytthe A, Moller S, Overgaard S, Brandt LP. Sex differences in risk and heritability estimates on primary knee osteoarthritis leading to total knee arthroplasty: a nationwide population based follow up study in Danish twins. Arthritis Res Ther. 2016 Feb 11;18:46. doi: 10.1186/s13075-016-0939-8. PMID 26864139
- [Background] Skousgaard SG, Hjelmborg J, Skytthe A, Brandt LP, Moller S, Overgaard S. Probability and heritability estimates on primary osteoarthritis of the hip leading to total hip arthroplasty: a nationwide population based follow-up study in Danish twins. Arthritis Res Ther. 2015 Nov 20;17:336. doi: 10.1186/s13075-015-0854-4. PMID 26589897
- [Derived] Heffernan SM, McCarthy C, Eustace S, FitzPatrick RE, Delahunt E, De Vito G. Mineral rich algae with pine bark improved pain, physical function and analgesic use in mild-knee joint osteoarthritis, compared to Glucosamine: A randomized controlled pilot trial. Complement Ther Med. 2020 May;50:102349. doi: 10.1016/j.ctim.2020.102349. Epub 2020 Feb 19. PMID 32444040
- See also: Algae-based food supplement PATENT — https://www.google.com/patents/EP1433388A1?cl=en
- See also: Method of preparing a novel antacid pharmaceutical product PATENT — https://www.google.com/patents/US3857938?dq=Rovati,+L.+(1972).&hl=en&sa=X&ved=0ahUKEwiRusGNtOfSAhVEDMAKHRhzDcYQ6AEIIDAB